CLINICAL TRIAL: NCT04662593
Title: Koa Family Study--A Community-Based Intervention to Improve Health and Well-Being
Acronym: KFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1668154
Record Dates: First submitted 2020-12-01; First posted 2020-12-10 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Overweight; Diet, Healthy; Social Interaction; Weight Loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group participates in a 17-week whole health program including:
  1. Weekly, small group online meetings with a health coach;
  2. Supportive social media including a private Facebook group and selective text messaging;
  3. Exposure to community tree planting and stewardship (through live streaming or in-person if COVID-19 public health guidance at the time, permits.
  Interventions: Behavioral: Whole Health Program
- Control Group (No Intervention): The control group participates only in questionnaire data collection at baseline, 4 months, and 6 months as well as daily weighing. Control group participants will be offered 3 web-based seminars (webinars) highlighting the effective lifestyle approaches demonstrated in the study and intervention group health education materials. The webinars and materials will be provided after the 6-month data collection which concludes the study.

INTERVENTIONS:
Behavioral: Whole Health Program — A mind-body-spirit intervention to improve health and well-being including weight loss.
  Arms: Intervention Group

SUMMARY:
Wholehearted living touches every aspect of life, from eating nourishing foods, to enjoying enough physical activity, to cultivating relationships that support healthy choices, to joining with neighbors to stand up for positive changes, and more. Unfortunately, for many low-income Californians, the idea of wholehearted living is an aspiration and not a reality. Koa Family: Strong, Healthy, Whole is an approach designed to make wholehearted living available for all.

The Approach Koa Family is a 4-month journey to establish "micro-communities" of women supporting one another- mind, body, and spirit. The foundation of this approach is a new, custom-designed, online Whole Health Program (WHP) that addresses healthy eating, physical activity, and weight management within the context of wholehearted living. Low-income women and a lifestyle coach will meet weekly in a virtual platform to learn, experience, grow, and thrive as they reach their diet, physical activity, and weight management goals.

Participants in the WHP will receive additional encouragement and access to local resources through a private and secure Facebook group. The group will provide a place for women to continue their wholehearted health journeys beyond the weekly meetings. Koa Family participants also will be invited to take part in a neighborhood tree planting campaign to create real, long-lasting, healthy changes to the environment in which they live.

The Study Koa Family, with WHP at its core, is the product of extensive formative research both nationally and within low-income California communities. Koa Family will be introduced in Sacramento County in February 2021. It will be evaluated for effectiveness among 120 low-income, Supplemental Nutrition Assistance Program (SNAP)-Ed eligible women using a randomized controlled trial study design, the gold standard for assessing effectiveness of an intervention. Outcomes include changes in Body Mass Index, diet, and physical activity measured at 4 and 6 months from baseline. An economic analysis will assess the cost-effectiveness of Koa Family, while qualitative methods will identify mediating factors related to the study outcomes.

Funding Koa Family is a project of the Population Health Group at the University of California, Davis, Center for Healthcare Policy and Research. Funding is provided by the United States Department of Agriculture Supplemental Nutrition Assistance Program-Education and the California Department of Forestry and Fire Protection (CalFIRE).

DETAILED DESCRIPTION:
The Koa Family Study is a randomized controlled trial testing a 17-week intervention, the Koa Family Program (KFP), consisting of three components: (1) the Whole Health Program (WHP)-a weekly, online group session facilitated by a health coach using the Zoom platform; (2) social media support including texting of health messages and a private Facebook group; and (3) a community empowerment arm designed around tree planting. The KFP addresses well-being from physical, mental, and social health perspectives. The program is intended to increase weight loss while fostering self-empowerment and connections to community resources to help sustain long-term weight management.

This study will test the following hypotheses:

1. Intervention participants, consisting of low-income overweight or obese women living in urban communities, receiving the KFP will have greater average weight loss and reduction in body mass index (BMI) than participants in the control group (who do not participate in the KFP);
2. KFP participants will show greater improvements in dietary practices compared with participants in the control group;
3. KFP participants will have greater increases in physical activity compared with control group participants;
4. KFP participants will have greater improvements in measures of well-being) compared with control group participants;
5. There will be a dose-response effect where greater engagement with the components of the KFP will be associated with larger improvements in the above endpoints (weight, diet, physical activity, and well-being).

Study design. The primary study will employ a prospective, randomized controlled trial (RCT) design. One hundred twenty eligible participants will be assigned to either the intervention (n=60) or control (n=60) group.

Intervention. The intervention group (n=60) will participate in the 17-week, KFP that supports physical, mental, and social well-being. It consists of: (1) theWHP-a weekly, online group session facilitated by a health coach using the Zoom platform; (2) social media support including texting of health messages and a private Facebook group; and (3) a community empowerment arm designed around tree planting.

The WHP is a small group-focused intervention designed to build "micro-communities" of mothers supporting one another in healthy living. Groups of 5-10 women living in the same community will meet online for 75 minutes weekly via the Zoom platform, for a total of 17 sessions. Each weekly session will cover a topic on whole-person living, including healthy eating, physical activity, weight management, coping, and resilience. The content of the WHP is based, in part, on the Centers for Disease Control and Prevention's National Diabetes Prevention Program (PT2) and Family Hui, a peer-led, women's group program to increase positive parenting skills and help families thrive.

For social media support, the intervention participants will receive brief text messages on their cell phones to encourage healthy lifestyle choices and connect to supportive community events and resources. EZTexting will be used to send text messages to participants. The participants also will be invited to join a private Facebook community, linked to each WHP group.

The principles and practice for tree planting and stewardship will be taught within the WHP sessions. If public health policy at the time, relating to managing Coronavirus Disease (COVID)-19 permits, participants may choose to participate in community tree plantings while complying with public health directives.

The control group participants will be enrolled for study measurements only and after the intervention period, will receive information based on what is proven effective in the RCT. This information will be delivered in a series of three webinars delivered after the last study data are collected at 25 weeks after baseline.

Data Collection. All participants will be asked to complete a phone-based, questionnaire administered by trained research staff. It will take about 50 minutes to complete the questionnaire. Questions will cover diet, physical activity, and well-being. The questionnaire will be administered at baseline, at week 18 after completion of the 17-week intervention, and at week 26 of the study.

At about week 8, an online focus group will be conducted as part of one of the sessions to qualitatively assess participants' experiences with the KFP.

Weight will be collected, daily, through a research-quality, Bluetooth-enabled scale that can transmit participant weights via the Internet to a secure server.

ELIGIBILITY:
Inclusion Criteria:

* female
* 21-45 years old
* comfortable speaking and reading English (all race/ethnicities are welcomed to participate)
* living in a low-income household (at or below 185% of the Federal Poverty Level)
* living in the Sacramento area
* familiarity with Facebook, Zoom, and texting
* access to a smartphone or high-speed internet (via a tablet or computer)
* overweight or obese (BMI≥25 and <39.9)

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* within 2 years postpartum;
* life-threatening illness;
* institutionalization (i.e., not free-living in the community);
* moderate to severe mental illness;
* receiving nutrition therapy from a health or health care provider (licensed or unlicensed);
* had or are considering bariatric surgery;
* medically diagnosed eating disorder;
* taking medication that affects weight;
* thyroid disease;
* Type 1 or Type 2 diabetes without medical clearance from the participant's physician;
* plans to move away during the study period.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 70 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Weight at 4 Months | Difference in weight between baseline and 4 months
  Weight (kg) measured with an electronic scale
Change from Baseline Weight at 6 Months | Difference in weight between baseline and 6 months
  Weight (kg) measured with an electronic scale
Change from Baseline Body Mass Index (BMI) at 4 Months | Difference in BMI between baseline and 4 months
  weight (kg)/height (m) x height (m)
Change from Baseline Body Mass Index (BMI) at 6 Months | Difference in BMI between baseline and 6 months
  weight (kg)/height (m) x height (m)
Change from Baseline Diet at 4 Months | Difference in diet between baseline and 4 months
  Measured with the Dietary Screener Questionnaire (NHANES 2009-10) to examine quality of participants' diet
Change from Baseline Diet at 6 Months | Difference in diet between baseline and 6 months
  Measured with the Dietary Screener Questionnaire (NHANES 2009-10) to examine quality of participants' diet
Change from Baseline Physical Activity (PA) at 4 Months | Difference in PA between baseline and 4 months
  Measured using the Centers for Disease Control and Prevention Behavioral Risk Factor Surveillance Survey Physical Activity Module
Change from Baseline Physical Activity (PA) at 6 Months | Difference in PA between baseline and 6 months
  Measured using the Centers for Disease Control and Prevention Behavioral Risk Factor Surveillance Survey Physical Activity Module
Change from Baseline Health-Related Well-being at 4 Months | Difference in health-related well-being between baseline and 4 months
  Well-being and general health measured with Short Form-36v2; There are 8 sections each scored 0-100 with a high score indicating less disability
Change from Baseline Health-Related Well-being at 6 Months | Difference in health-related well-being between baseline and 6 months
  Well-being and general health measured with Short Form-36v2

CONTACTS AND LOCATIONS:
Overall Officials: Desiree Backman, DrPH, MS, RD, Principal Investigator — UC Davis Center for Healthcare Policy and Research
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA. 2012 Feb 1;307(5):491-7. doi: 10.1001/jama.2012.39. Epub 2012 Jan 17. PMID 22253363
- [Background] Abdelaal M, le Roux CW, Docherty NG. Morbidity and mortality associated with obesity. Ann Transl Med. 2017 Apr;5(7):161. doi: 10.21037/atm.2017.03.107. PMID 28480197